CLINICAL TRIAL: NCT00065143
Title: A Phase II Study of Clofarabine in Combination With Cytarabine (Ara-C) in Patients >/= 50 Years With Newly Diagnosed and Previously Untreated Acute Myeloid Leukemia (AML) and High-risk Myelodysplastic Syndrome (MDS) (>/= 10% Bone Marrow Blasts)
Brief Title: Clofarabine Plus Cytarabine in Patients With Previously Untreated Acute Myeloid Leukemia and High-risk Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID03-0139
Record Dates: First submitted 2003-07-17; First posted 2003-07-18 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Leukemia, Myeloid; Myelodysplastic Syndromes
Keywords: Newly diagnosed and previously untreated acute myeloid leukemia (AML); High-risk myelodysplastic syndrome (MDS) (>/= 10% bone marrow blasts); Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS)
MeSH Terms: conditions — Leukemia, Myeloid; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Clofarabine; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: clofarabine
Drug: Ara-C

SUMMARY:
The goal of this clinical research study is to learn if clofarabine, when given in combination with ara-C (cytarabine), can help to improve the disease's response to therapy and to increase the duration of response in patients who are 50 years or older with leukemia. The safety of this combination treatment will also be studied.

DETAILED DESCRIPTION:
The treatment of acute myeloid leukemia (AML) in older patients has not improved significantly in recent years when compared with the considerable progress that has been made in younger patients. Hence, new drugs and approaches are needed in this poor-prognosis group of patients with AML.

Nucleoside analogs are among the most active antileukemic agents available. Clofarabine was synthesized as a rational extension of the experience with other deoxyadenosine analogs. Clofarabine is converted to the monophosphate form by the enzyme deoxycytidine kinase which represents the major metabolite of clofarabine. Phosphorylation of clofarabine is substantially more efficient than that of other nucleosides such as fludarabine and so is intracellular retention of the triphosphate form of clofarabine. Mechanisms of action include inhibition of DNA synthesis, inhibition of DNA polymerases, and potent inhibition of ribonucleotide reductase (RNR) resulting in depletion of normal nucleotides and increased DNA uptake of the analog. Single agent clofarabine has shown activity in phase I studies in AML and ALL. As a potent inhibitor of RNR, however, clofarabine is ideal to be incorporated into biochemical modulation strategies such as have been tested and validated with fludarabine and ara-C in AML. By combining clofarabine with ara-C, inhibition of RNR by clofarabine will result in a drop of deoxynucleotides causing a decrease in the feedback inhibition of deoxycytidine kinase which is the rate-limiting step in the synthesis of ara-CTP leading to increased retention of ara-CTP. Therefore, the activity of clofarabine and ara-C in leukemic cells would be complemented by a biochemical synergism between these agents that should result in better clinical efficacy. We have established the safety of the combination in salvage patients with acute leukemias.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated acute myeloid leukemia (AML) or high-risk myelodysplastic syndrome (MDS) (> 10% blasts). Prior therapy with hydroxyurea, single agent chemotherapy (e.g. decitabine), hematopoietic growth factors, biological or "targeted" therapies are allowed.
* Age > 50 years to < 74 years (diploid cytogenetics) and < 69 years (abnormal cytogenetics).
* ECOG performance status </= 2.
* Sign a written informed consent form.
* Adequate liver function (total bilirubin < 2mg/dL, SGPT or SGOT < x 4 ULN) and renal function (serum creatinine < 2mg/dL).
* Male and female patients who are fertile agree to use an effective barrier method of birth control (ie, latex condom, diaphragm, cervical cap, etc) to avoid pregnancy. Female patients need a negative serum or urine pregnancy test within 7 days of study enrollment (applies only if patient is of childbearing potential. Non-childbearing is defined as >= 1 year postmenopausal or surgically sterilized).
* Patients who are considered to require immediate induction (rapidly rising WBC >/= 50,000 and/or organ involvement as per the assessment of the treating physician) can be treated without final cytogenetic results and pretreatment assessment of cardiac ejection fraction (MUGA or echocardiogram) if by history and physical examination patients have </= NYHA class II disease.

Exclusion Criteria:

* AML with the following cytogenetic abnormalities: t(15;17), t(8;21), inv(16). Cytogenetic results do not need to be available if immediate induction is required (see inclusion #7).
* Cardiac ejection fraction < 30%. Pretreatment assessment of ejection fraction is not necessary if immediate induction is required as long as by history and physical examination patients have </= NYHA class II disease (see inclusion #7).
* Active and uncontrolled infection or any other severe concurrent disease considered life-threatening, or which, in the judgement of the investigator and after discussion with the Principal Investigator, would make the patient inappropriate for entry into the study.

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2003-06-23 (Actual); Primary Completion 2006-02-22 (Actual); Study Completion 2006-02-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Faderl, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: Website for The University of Texas M.D. Anderson Cancer Center — http://www.mdanderson.org